CLINICAL TRIAL: NCT06436105
Title: Comparison of Perioperative Analgesic Effectiveness of Patients Who Had Fasia Iliac Compartment Block and 4in1 Block Applied in Total Knee Prosthesis Surgery
Brief Title: Comparison of Fasia Iliac Compartment Block and 4in1 Block
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Diskapi Yildirim Beyazit Education and Research Hospital (Other Government)
Responsible Party: Principal Investigator, Savas Altinsoy, Principal Investigator, Diskapi Yildirim Beyazit Education and Research Hospital
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Other
Other Study IDs: İsa Öteleş
Record Dates: First submitted 2024-05-24; First posted 2024-05-30 (Actual); Last update posted 2025-06-29 (Actual); Status verified 2025-06

CONDITIONS: Pain, Postoperative
Keywords: FICB; 4 in 1 block; Total knee arthroplasty
MeSH Terms: conditions — Pain, Postoperative

STUDY DESIGN:
Who Masked: Participant
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (3):
- Group Control (Other): Peripheral nerve block will not be performed on Group Control patients.
  Interventions: Other: Control
- Group FICB (Other): FICB will be performed with 30 ml %0.25 bupivacaine for Group FICB patients.
  Interventions: Other: FICB
- Group 4 IN 1 (Other): 4 in 1 block will be performed with 30 ml %0.25 bupivacaine for Group 4 IN 1 patients.
  Interventions: Other: 4 in 1 block

INTERVENTIONS:
Other: FICB — FICB is applied to the patients after spinal anesthesia.
  Arms: Group FICB
Other: 4 in 1 block — 4 in 1 block is applied to the patients after spinal anesthesia.
  Arms: Group 4 IN 1
Other: Control — Peripheral nerve block will not be performed on Group Control patients.
  Arms: Group Control

SUMMARY:
Patients who will undergo elective total knee arthroplasty surgery under spinal anesthesia will be included in the study according to the postoperative analgesia method applied: Group Control, Group FICB and Group 4in1. Peripheral nerve block will be performed with 30 ml %0.25 bupivacaine for Group FICB and Group 4 in 1 patients. Peripheral nerve block will not be performed on Group Control patients. Patient-controlled analgesia will be given to all three groups in the postoperative period. PCA is a pain palliation method routinely used in all patients postoperatively. NRS score, PCA tramadol consumption, PCA demand, need for additional analgesia, patient satisfaction, nausea and vomiting will be monitored 24 hours postoperatively. The aim of this study is to compare the perioperative analgesic effectiveness of patients who underwent fascia iliaca compartment block and 4 in 1 block in total knee arthroplasty surgery, with each other and with the control group.

DETAILED DESCRIPTION:
Total knee arthroplasty is a surgical procedure performed mostly on patients with osteoarthritis who have failed traditional conservative treatment. Increasing knee osteoarthritis due to reasons such as life expectancy and body mass index causes this surgical procedure to be performed more frequently. The knee joint which is innervated by the femoral, obturator, sciatic nerves and their branches has a complicated innervation and the pain following total knee arthrplasty is quite severe. It is aimed to provide effective analgesia by blocking these nerves or terminal branches with various peripheral nerve blockade methods under USG guidance. In recent years, interest in studies aiming to block these nerves with a single injection has been increasing. 4 in 1 block is a new technique applied from a single injection point to block the saphenous, obturator, sciatic and vastus medialis nerves that innervate the knee joint. Fascia iliaca compartment block is a reliable technique applied from a single injection point to block the femoral, lateral femoral cutaneous and obturator nerves behind the fascia iliaca.

Patients who will undergo elective total knee arthroplasty surgery under spinal anesthesia will be included in the study according to the postoperative analgesia method applied: Group Control, Group FICB and Group 4in1. Peripheral nerve block will be performed with 30 ml %0.25 bupivacaine for Group FICB and Group 4 in 1 patients. Peripheral nerve block will not be performed on Group Control patients. Patient-controlled analgesia will be given to all three groups in the postoperative period. PCA is a pain palliation method routinely used in all patients postoperatively. NRS score, PCA tramadol consumption, PCA demand, need for additional analgesia, patient satisfaction, nausea and vomiting will be monitored 24 hours postoperatively. The aim of this study is to compare the perioperative analgesic effectiveness of patients who underwent fascia iliaca compartment block and 4 in 1 block in total knee arthroplasty surgery, with each other and with the control group.

ELIGIBILITY:
Inclusion Criteria:

* With informed consent
* Elective total knee arthroplasty with spinal anesthesia
* Oriented and cooperative
* ASA Classification I-II-III
* 18-85 years old

Exclusion Criteria:

* Anticoagulant medication
* Coagulopathy
* Infection at the site of peripheral nerve block application
* Allergy to local anesthetics
* Pregnant or suspected pregnancy

Ages: 18 Years to 85 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 60 (Actual)
Dates: Start 2024-05-30 (Actual); Primary Completion 2024-07-01 (Actual); Study Completion 2024-07-08 (Actual)

PRIMARY OUTCOMES:
Total tramadol consumption in 24 hours (mg) | 24 hours postoperatively
  Total tramadol consumption used in the first 24 hours postoperatively

SECONDARY OUTCOMES:
Pain on the Numeric Rating Scale (NRS) | 0 hours postoperatively
  NRS range was from 0-10 with being no pain and 10 the worst pain possible.
Pain on the Numeric Rating Scale (NRS) | 1 hours postoperatively
  NRS range was from 0-10 with being no pain and 10 the worst pain possible.
Pain on the Numeric Rating Scale (NRS) | 4 hours postoperatively
  NRS range was from 0-10 with being no pain and 10 the worst pain possible.
Pain on the Numeric Rating Scale (NRS) | 8 hours postoperatively
  NRS range was from 0-10 with being no pain and 10 the worst pain possible.
Pain on the Numeric Rating Scale (NRS) | 12 hours postoperatively
  NRS range was from 0-10 with being no pain and 10 the worst pain possible.
Pain on the Numeric Rating Scale (NRS) | 24 hours postoperatively
  NRS range was from 0-10 with being no pain and 10 the worst pain possible.
Rescue Analgesic | 24 hours postoperatively
  Consumption of rescue analgesic used after 24 hours postoperatively.
Patient satisfaction | 24 hours postoperatively
  The patient is satisfied or dissatisfied

CONTACTS AND LOCATIONS:
Locations (1):
- Department of Anesthesiology and Reanimation, University of Health Sciences, Diskapi Yıldırım Beyazit Training and Research Hospital, Ankara, Turkey (Türkiye)

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] Roy R, Agarwal G, Pradhan C, Kuanardr D, Mallick DJ. Ultrasound guided 4 in 1 block - a newer, single injection technique for complete postoperative analgesia for knee and below knee surgeries. Anaesthesia, Pain & Intensive Care. 2018;22(1):87-92.
- [Result] Kanadli H, Dogru S, Karaman T, Karaman S, Tapar H, Sahin A, Asci M, Kanadli KA, Suren M. Comparison of the efficacy of femoral nerve block and fascia iliaca compartment block in patients with total knee replacement. Minerva Anestesiol. 2018 Oct;84(10):1134-1141. doi: 10.23736/S0375-9393.18.12062-1. Epub 2018 Jan 16. PMID 29338141